CLINICAL TRIAL: NCT06451614
Title: SpaceIT Hydrogel System for Perirectal Spacing in Subjects With Low to Intermediate Risk Prostate Cancer Undergoing External Beam Radiotherapy (EBRT)
Brief Title: SpaceIT Hydrogel System for Perirectal Spacing
Acronym: HYDROSPACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U0755
Record Dates: First submitted 2024-05-07; First posted 2024-06-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- SpaceIT Hydrogel System (Experimental): Subjects randomized to the investigational arm will undergo a hydrogel procedure with the SpaceIT investigational device.
  Interventions: Device: SpaceIT Hydrogel System
- Commercially available Boston Scientific Spacer (Active Comparator): Subjects randomized to the control arm will undergo a hydrogel procedure with the Boston Scientific commercially available SpaceOAR or SpaceOAR VUE device.
  Interventions: Device: Commercially available Boston Scientific Spacer

INTERVENTIONS:
Device: SpaceIT Hydrogel System — SpaceIT Hydrogel System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer and in creating this space it is the intent of SpaceIT Hydrogel System to reduce the radiation dose delivered to the anterior rectum. The SpaceIT Hydrogel System is composed of a radiopaque, biodegradable material designed to maintain space for approximately 12 weeks and be absorbed in about 6 months, sufficient time to support the intended use.
  SpaceIT has an iodinated PEG powder making it radiopaque.
  Arms: SpaceIT Hydrogel System
Device: Commercially available Boston Scientific Spacer — Boston Scientific's commercially available SpaceOAR Hydrogel System or SpaceOAR Vue Hydrogel System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer and in creating this space it is the intent of SpaceOAR Hydrogel System or SpaceOAR Vue Hydrogel System to reduce the radiation dose delivered to the anterior rectum. SpaceOAR and SpaceOAR Vue are both perirectal spacers. SpaceOAR Vue specifically has an iodinated PEG powder making it radiopaque. SpaceOAR does not contain iodinated PEG powder and is not radiopaque. The SpaceOAR Hydrogel System or SpaceOAR Vue Hydrogel System maintains space during prostate radiotherapy treatment and is completely absorbed by the patient's body over time.
  Arms: Commercially available Boston Scientific Spacer

SUMMARY:
To evaluate the safety and effectiveness of the SpaceIT™ Hydrogel System in patients undergoing External Beam Radiotherapy (EBRT) for the treatment of prostate cancer.

DETAILED DESCRIPTION:
HYDROSPACE study is a prospective, randomized, multicenter study to evaluate the safety and effectiveness of SpaceIT in patients undergoing External Beam Radiotherapy (EBRT) for the treatment of prostate cancer.

Subjects randomized to the investigational arm will receive SpaceIT Hydrogel System

Subjects randomized to the control arm will receive a commercially marketed Boston Scientific perirectal hydrogel spacer, SpaceOAR System or SpaceOAR Vue Hydrogel

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for participation in the study:

1. Age ≥18 years old
2. Subjects must have had pathologically confirmed (by routine hematoxylin and eosin [H&E] staining) invasive adenocarcinoma of the prostate and planning to undergo EBRT
3. Subjects must meet ALL of the following:

   1. Clinical stage T1-T2c (AJCC Ver. 8) tumor AND
   2. Gleason Score 7 or less as determined from a biopsy taken within 12 months of the Baseline visit AND
   3. Demonstrated blood prostate specific antigen (PSA) levels ≤20 ng/ml as measured within 6 months of the Baseline visit and prior to commencing androgen deprivation therapy (ADT)
4. Subject is able to provide written informed consent, approved by the appropriate Institutional Review Board/Ethics Committee/Research Ethics Board (IRB/EC/REB) of the respective clinical site

Exclusion Criteria:

1. Prostate > 80 cc
2. Subjects who are planning to undergo brachytherapy or focal boost
3. Subjects who have magnetic resonance imaging (MRI) evidence of gross posterior extracapsular extension (ECE) of the prostate cancer Note: MRI must be taken within 6 months prior to the Baseline visit
4. Subjects who have metastatic disease, other ongoing cancers which are being treated during the study or subjects for whom pelvic lymph node radiotherapy is planned
5. Subjects with any prior invasive solid tumor malignancy or hematologic malignancy (except non-melanomatous skin cancer) unless the subject has been disease free and treatment free for a minimum of 3 years
6. History of radical prostatectomy, other ablative anti-prostate cancer therapy (e.g., cryotherapy, high intensity focused ultrasound, irreversible electroporation) or previous pelvic irradiation (including prior prostate brachytherapy) at any time prior to screening
7. History of transurethral prostate surgery (e.g., Transurethral Needle Ablation (TUNA), Transurethral Microwave Therapy (TUMT), Transurethral Resection of the Prostate (TURP)) if performed within 1 year prior to screening
8. History of prior pelvic surgery requiring low anterior or abdominoperineal resections or rectal surgery
9. History of or current perirectal disease that may interfere with interpretation of study outcomes, including anal or perianal diseases such as fistula
10. Bleeding hemorrhoids requiring medical intervention within the prior three months
11. Diagnosed active bleeding disorder or a clinically significant coagulopathy, defined as PTT > 70s or aPTT>35s or INR > 1.4, or platelet count < 100,000 per mm3 Note: Subjects on anticoagulants may be included if the anticoagulant medication can be held for index procedure
12. Active inflammatory or infectious process involving the perineum, GI or urinary tract based on positive diagnosis or suspected diagnosis in the presence of fever >38⁰ C, WBC > 12,000/uL
13. Inability to undergo pelvic MRI or presence of implants causing severe artifact (e.g. bilateral arthroplasty) that interferes with imaging interpretation for this study at Investigator discretion
14. If a subject was enrolled in another investigational drug or device trial that had not completed the primary endpoint or that clinically interfered with this study
15. Unable to comply with the study requirements or follow-up schedule
16. Any condition the Investigator believed would interfere with the intent of the study or would make participation not in the best interest of the patient
17. Known PEG (polyethylene glycol) sensitivity or allergy
18. Known iodine sensitivity or allergy
19. ADT, if applicable, cannot or was not started 15-60 days prior to the pre-index procedure RT planning imaging and is planned to continue for a total planned duration greater than 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 230 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Acute Grade 3 or greater adverse events. | 90 Days from hydrogel placement procedure
  Acute Grade 3 or greater adverse events, inclusive of all adverse events listed on the existing SpaceOAR product labels, that arise within 90 days of index procedure.
Primary Effectiveness Endpoint - 25% reduction in the volume of the rectum receiving 90% of the prescribed radiation dose | 10 days post procedure
  Clinically relevant dose reduction defined as a 25% reduction in the volume of the rectum receiving 90% of the prescribed radiation dose in subjects receiving hydrogel.

SECONDARY OUTCOMES:
Additional Safety Endpoint - Adverse Device Effects (ADEs) requiring additional procedures and/or medications | Up to 24 months
  Adverse Device Effects (ADEs) requiring additional procedures and/or medications
Additional Safety Endpoint - Incidence of acute Grade 2 or greater gastrointestinal (GI) and genitourinary (GU) adverse events (AEs) | Up to 90 days
  Incidence of acute Grade 2 or greater gastrointestinal (GI) and genitourinary (GU) adverse events (AEs) from index procedure up to 3 months
Additional Safety Endpoint - Incidence of late Grade 2 or greater GI and GU adverse events (AEs) | 91 days up to 24 Months
  Incidence of late Grade 2 or greater GI and GU adverse events (AEs) from 3 months up to the end of study follow-up
Additional Effectiveness Endpoint - Visualization of hydrogel | 10 days post procedure
  Technical Success: visualization of hydrogel between the posterior prostatic capsule and the anterior rectal wall will be assessed as Yes/No using the MRI performed post hydrogel placement procedure
Additional Effectiveness Endpoint - Space Creation | 10 days post procedure
  Space Creation: Distance between the posterior prostatic capsule and anterior rectal wall will be measured mid gland in millimeters using MRI performed post hydrogel placement procedure
Additional Effectiveness Endpoint - Absorption | 12 Month post hydrogel placement
  Absorption: Absence of hydrogel in the perirectal space assessed on MRI at 12 months post-hydrogel placement.
Additional Effectiveness Endpoint - Change in radiation dose distributions to the organs at risk | 10 days post procedure
  Dose Distribution: Change in radiation dose distributions to the organs at risk (OARs) quantified by computing rectal Dose-Volume Histograms (DVHs) for the dose plans created pre-and post-hydrogel placement.
Additional Effectiveness Endpoint - Mean and Maximum Rectal Radiation doses | 10 days post procedure
  Mean and Maximum Rectal Radiation Doses (in Gy)
Additional Effectiveness Endpoint - Quality of Life Questionnaire: EQ-5D-5L | Baseline up to 24 months
  Changes from Baseline in EQ-5D-5L
  The EQ-5D-5L is a generic questionnaire that assesses a subject's self-reported health status in terms of five dimensions of health: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Subject's overall current health on a vertical visual analogue scale of "0-100" is recorded, where the endpoints are labelled 'The best health you can imagine' at "100" and 'The worst health you can imagine' at "0".
Additional Effectiveness Endpoint - Ease of hydrogel administration | 10 days post procedure
  Ease of hydrogel administration. Scored on a Likert scale from 1 to 5 where 1 is Very Difficult and 5 is Very Easy
Additional Effectiveness Endpoint - Space Maintenance | 3 Months post hydrogel placement procedure
  Space Maintenance: Distance between the posterior prostatic capsule and anterior rectal wall will be measured
Additional Effectiveness Endpoint - Quality of Life Questionnaire: Expanded Prostate Cancer Index Composite (EPIC-26) | Baseline up to 24 months
  Changes from Baseline in Expanded Prostate Cancer Index Composite (EPIC-26)
  EPIC-26 is a questionnaire designed to measure health related quality of life (HRQOL) in people with prostate cancer. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Additional Effectiveness Endpoint - Quality of Life Questionnaire, Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) | Baseline up to 24 months
  Changes from Baseline in Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH)
  The Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Baumann, MD, Principal Investigator — Springfield Clinic
Locations (29):
- United States (26):
  - City of Hope, Duarte, California
  - Orange County Urology Associates, Laguna Hills, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Baptist Hospital of Miami, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - UroPartners, Glenview, Illinois
  - Springfield Clinic, LLC, Springfield, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Integrated Medical Professionals, New York, New York
  - Perlmutter Cancer Center - NYU Langone, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Northwell Health, New York, New York
  - University Hospitals of Cleveland-Hospital, Cleveland, Ohio
  - Mercy Cancer Center Bon Secours Mercy Healt, Elyria, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Gibbs Cancer Center and Research Institute, Greer, South Carolina
  - Midtown Urology Associates, Austin, Texas
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - Rio Grande Urology, El Paso, Texas
  - Houston Metro Urology, Houston, Texas
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - University of Washington Medical Center-Hospital, Seattle, Washington
- Canada (3):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre-Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No